CLINICAL TRIAL: NCT05287906
Title: The Effects of Steviol Glycosides on Acute Appetite Hormone Release in Men and Women with Normal Weight, Overweight and Type 2 Diabetes
Brief Title: A Trial to Assess Steviol Glycosides on Acute Appetite Hormone Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Center for Metabolic and Cardiovascular Research (Other)
Collaborators: Cargill (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MB-2110
Record Dates: First submitted 2022-03-10; First posted 2022-03-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Overweight and Obesity; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2 | interventions — Water; Glucose; rebaudioside A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Normal Weight Group (Experimental): The normal weight group incudes men and women with BMI 18.5 - 24.9 kg/m2, and will receive all interventions.
  Interventions: Other: Water; Other: Glucose; Other: Steviol Glycosides; Other: Steviol Glycosides plus glucose; Other: Rebaudioside A
- Overweight Group (Experimental): The overweight group includes men and women with BMI 25.0 - 29.9 kg/m2, and will receive all interventions.
  Interventions: Other: Water; Other: Glucose; Other: Steviol Glycosides; Other: Steviol Glycosides plus glucose
- Type 2 Diabetes Mellitis Group (Experimental): The T2DM group includes men and women with BMI 25.0 - 34.9 kg/m2, HbA1c <8%, and will receive all interventions.
  Interventions: Other: Water; Other: Glucose; Other: Steviol Glycosides; Other: Steviol Glycosides plus glucose

INTERVENTIONS:
Other: Water — Each subject will receive one control and three treatments in the crossover design. The control contains water only.
Other: Glucose — Each subject will receive one control and three treatments in the crossover design. The glucose contains water and glucose.
Other: Steviol Glycosides — Each subject will receive one control and three treatments in the crossover design. The Steviol Glycoside beverage contains water and steviol glycosides.
Other: Steviol Glycosides plus glucose — Each subject will receive one control and three treatments in the crossover design. The Steviol Glycoside plus glucose beverage contains water, glucose, and steviol glycosides.
Other: Rebaudioside A — A leaf-based, extracted stevia product to compare to the Eversweet in the normal weight group only. The Rebaudioside A contains water and rebaudioside A.
  Arms: Normal Weight Group

SUMMARY:
The objectives of this trial are to assess the effects of steviol glycoside alone or in combination with a glycemic carbohydrate on blood glucose and endocrine and gut hormone secretion vs. water and glucose in individuals with normal weight, overweight and type 2 diabetes mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female and is 18-50 years of age, inclusive.
2. Subject has BMI 18.5 to 24.9 kg/m2, inclusive, for the normal weight group.
3. Subject has BMI 25.0 to 29.9 kg/m2, inclusive, for the overweight group.
4. Subject has BMI 25.0 to 34.9 kg/m2, inclusive, and HbA1c <8%, and is not taking any injectable hypoglycemic medication(s) or oral glucagon-like peptide 1 (GLP-1) mimetic(s), for individuals with T2DM.
5. Subject has consumed ≤670 mL (24 oz) of artificially sweetened or steviol glycoside sweetened soft drinks per week for at least 1 month before screening.
6. Consumption of less than 2 yogurts per week (that are sweetened with HIS).
7. Subject has a score of at least 7 on the Vein Access Scale.
8. Subject is willing to follow his/her regular physical activity pattern throughout the study period.
9. Subject is willing to refrain from consuming marijuana throughout the study period.
10. Subject is willing to refrain from consumption of alcoholic beverages for 48 h prior to each clinic visit.
11. Subject is willing to refrain from vigorous physical activity for 24 h prior to each clinic visit. According to the World Health Organization (WHO), vigorous physical activity may include running, fast cycling, fast swimming, or moving heavy objects.
12. Subject is willing to abstain from tobacco use 1 h prior to and during each clinic visit and has no plans to change smoking, vaping or other nicotine use habits during the study period
13. Subject understands the study procedures and is willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study Investigator.

Exclusion Criteria:

1. Subject has a laboratory test result of clinical significance in the opinion of the study Investigator at visit 1 (week -1).
2. Subject has atherosclerotic cardiovascular disease including any of the following: clinical signs of atherosclerosis including peripheral arterial disease, abdominal aortic aneurysm, carotid artery disease [symptomatic (e.g., myocardial infarction, angina, transient ischemic attack or stroke of carotid origin) or >50% stenosis on angiography or ultrasound] or other forms of clinical atherosclerotic disease (e.g., renal artery disease).
3. Subject has a history or presence of a clinically important medical condition that, in the opinion of the Investigator, could interfere with the interpretation of the study results.
4. Individual has a positive urine drug screen for illicit drugs.
5. Individual has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg and/or diastolic blood pressure ≥100 mm Hg) at visit 1 (week -1).
6. Subject has a history of cancer in the prior 5 years, except for non-melanoma skin cancer or carcinoma in situ of the cervix.
7. Subject has history of moderate or severe renal failure, moderate or severe liver disease, gall bladder removal, pancreatic disease, or a gastrointestinal disorder that might influence the digestion or absorption of nutrients or impact colonic function as judged by the Investigator.
8. Subject has history of major trauma or a major medical or surgical event requiring hospitalization within 3 months of visit 1 (week -1).
9. Subject has used antibiotics within 4 weeks of visit 1 (week -1) or has a condition likely to require the use of antibiotics during the study.
10. Subject has an active infection or has used antibiotics within 7 d of any test visit. Those with an active infection and/or using antibiotics must wait at least 7 d after the infection resolves or antibiotic use is complete. The test period will be extended for completion in these cases.
11. Subject has experienced a change in body weight of ±4.5 kg (~10 pounds) over the 3 months prior to visit 1 (week -1).
12. Subject has unstable use (initiation or dose alteration) of any antihypertensive medication within 4 weeks prior to visit 1 (week -1).
13. Subject has unstable use (initiation or dose alteration) of any of the following lipid-altering medications within 4 weeks prior to visit 1 (week -1): statins, ezetimibe, bempedoic acid, bile acid sequestrants, fibrates, niacin (drug form), and/or omega-3 fatty acid drugs.
14. Subject has unstable use (initiation or dose alteration) of a proprotein convertase subtilisin kexin type 9 (PCSK9) inhibitor within 3 months of visit 1 (week -1).
15. Subject has used weight-loss drugs (including over-the-counter medications and/or supplements) within 4 weeks of visit 1 (week -1).
16. Subject has used or has a condition likely to require the use of systemic corticosteroid drugs within 4 weeks of visit 1 (week -1).
17. Subject has unstable use (initiation or dose alteration) of medications known to influence carbohydrate metabolism, including, but not limited to, adrenergic receptor blockers, thiazide diuretics, hypoglycemic medications, and/or antipsychotics within 4 weeks prior to visit 1 (week -1).
18. Subject has used cannabidiol (CBD) products within two weeks prior to visit 2 (week 0) and throughout the study.
19. Subject has a known allergy, sensitivity, or intolerance to any ingredients in the study beverages.
20. Subject is a female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and unwilling to commit to the use of a medically approved form of contraception throughout the study period.
21. Subject has extreme dietary habits (e.g., vegan or very low carbohydrate diet).
22. Subject has a current or recent history (past 12 months), or strong potential, for drug or alcohol abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1 ½ oz distilled spirits).
23. Subject has a history of a diagnosed eating disorder (e.g., anorexia nervosa or bulimia nervosa).
24. Subject has been exposed to any non-registered drug product within 30 d of visit 1 (week -1).
25. Subject has a condition the Investigator believes would interfere with his or her ability to provide informed consent or comply with the study protocol, or which might confound the interpretation of the study results or put the person at undue risk.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Insulin | 4 weeks
  Changes or percent changes from baseline to the end of treatment
Glucose | 4 weeks
  Changes or percent changes from baseline to the end of treatment
Glucagon | 4 weeks
  Changes or percent changes from baseline to the end of treatment
Peptide YY | 4 weeks
  Changes or percent changes from baseline to the end of treatment
Glucagon-like peptide 1 | 4 weeks
  Changes or percent changes from baseline to the end of treatment
Gastric inhibitory polypeptide | 4 weeks
  Changes or percent changes from baseline to the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Maki, PhD, Study Director — MB Clinical Research & Consulting, LLC
Locations (3):
- United States (3):
  - Excellence Medical and Research, Miami Gardens, Florida
  - Advanced Research for Health Improvement, Naples, Florida
  - Great Lakes Clinical Trials, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No